CLINICAL TRIAL: NCT00414960
Title: Phase IIB Randomized, Placebo-Controlled, Double-Blind Study of Enzastaurin HCL (LY317615) for Lung Cancer Prevention in Former Smokers
Brief Title: A Trial of Placebo Versus Enzastaurin for Lung Cancer Prevention in Former Smokers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 10723; H6Q-MC-S009 (Other: Eli Lilly and Company); NCT00387816 (obsolete NCT alias)
Record Dates: First submitted 2006-12-21; First posted 2006-12-22 (Estimated); Results first posted 2020-09-21 (Actual); Last update posted 2020-09-21 (Actual); Status verified 2020-08

CONDITIONS: Lung Cancer
Keywords: Healthy; Prevention
MeSH Terms: conditions — Lung Neoplasms | interventions — enzastaurin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Enzastaurin (Experimental): Treatment with enzastaurin 500 milligrams (mg) orally (po) once daily (QD) given as 4 tablets (125 mg each).
  Interventions: Drug: Enzastaurin
- Placebo (Placebo Comparator): Treatment with placebo po QD appearing identical to enzastaurin.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Enzastaurin — 500 mg po QD for 6 months
  Other Names: LY317615
  Arms: Enzastaurin
Drug: Placebo — po QD for 6 months
  Arms: Placebo

SUMMARY:
To compare the difference of a marker of cellular proliferation in all bronchial biopsy specimens of former smokers stratified by lung cancer risk, collected before and after treatment per patient between the enzastaurin and placebo groups.

ELIGIBILITY:
Inclusion Criteria:

* Sputum atypia participants with normal sputum cytology will be removed from the study)
* Metaplasia or dysplasia on at least one bronchoscopy specimen
* History of cigarette smoking ≥30 Pack Years
* Quit smoking ≥1 year prior to study entry
* Able to undergo bronchoscopy and helical computed tomography (CT) scanning of the chest
* Able to swallow tablets

Exclusion Criteria:

* Blood clotting abnormalities
* Current smoking within the past 1 year
* Unwillingness to abstain from smoking while enrolled in the clinical trial or unwillingness to avoid significant second hand smoke exposure
* Evidence for lung cancer or carcinoma in situ
* Active cardiovascular disease
* Current illicit drug or alcohol abuse

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2007-12; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tampa, Florida, United States

REFERENCES:
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Enzastaurin: Treatment with enzastaurin 500 milligrams (mg) orally (po), once daily (QD) given as 4 tablets (125 mg each).
Period: Overall Study
Arm/Group | Enzastaurin | Placebo
Started | 25 | 15
Received at Least One Dose of Study Drug | 24 | 15
Completed | 18 | 14
Not Completed | 7 | 1
Not completed — Adverse Event | 4 | 0
Not completed — Withdrawal by Subject | 3 | 0
Not completed — Physician Decision | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Enzastaurin | Placebo | Total
Number analyzed (Participants) | 25 | 15 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.84 (6.06) | 66.97 (4.67) | 66.89 (5.51)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 8 | 14
  Male | 19 | 7 | 26
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 24 | 15 | 39
  Hispanic | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 25 | 15 | 40
Evidence of Airway Obstruction [Count of Participants; unit: Participants] — Evidence of airway obstruction present if Forced Expiratory Volume in 1 second/Forced Vital Capacity (FEV1/FVC ratio) ≤0.7; evidence of airway obstruction absent if FEV1/FVC ratio >0.7.
  Participants
    Absence | 13 | 11 | 24
    Presence | 12 | 4 | 16
Eastern Cooperative Oncology Group (ECOG) [Count of Participants; unit: Participants] — Measure of performance status as defined by ECOG on a scale of Grade 0 to Grade 5: 0=Fully active, able to carry on pre-disease performance without restriction; 1=Restricted in physically strenuous activity but ambulatory and able to carry out light and sedentary work; 2=Ambulatory and capable of all self-care but unable to carry out any work activities. Up and about more than 50% of waking hours; 3=Capable of only limited self-care, confined to bed or chair more than 50% of waking hours; 4=Completely disabled. Cannot carry on any self-care. Totally confined to bed or chair; 5=Dead.
  Participants
    Grade 0 | 19 | 12 | 31
    Grade 1 | 6 | 3 | 9
History of Stage I Non-small Cell Lung Cancer [Count of Participants; unit: Participants] — Participants were asked if they have a history of Stage 1 (cancer is small and has not spread to the lymph nodes) Non-small Cell Lung Cancer.
  Participants
    Yes | 1 | 1 | 2
    No | 24 | 14 | 38

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Percentage of Cells Staining Positive for Ki-67 in All Biopsy Specimens at Endpoint
Description: The number of cells positively stained for Ki-67 (a marker of cellular proliferation) was enumerated and divided by the total number of cells in each specimen. The average Ki-67 labeling index (LI) (percentage of cells positively labeled with Ki-67) for all histological specimens was then calculated for each participant.
Time Frame: Baseline, endpoint (up to 8 months)
Population: The number of participants analyzed was based on the efficacy population (EP). The EP included participants who met study criteria, were randomized to the study, and who had Ki-67 measurements from biopsy specimens.
Measure: Mean (Standard Deviation); unit: percentage of cells with Ki-67
Arm/Group | Enzastaurin | Placebo
Number analyzed (Participants) | 21 | 13
percentage of cells with Ki-67 | 3.74 (11.68) | 6.15 (11.08)
Statistical Analysis 1: Comparison: Enzastaurin vs Placebo; Test type: Superiority or Other; p = 0.556, 2-sample pooled t-test — P-value is for comparison of change from baseline between enzastaurin and placebo group; Mean Difference (Final Values) = -2.40, 95% CI 2-sided [-10.64 to 5.83], Standard Error of Mean 4.04 — Using placebo as a reference group, the mean difference = enzastaurin minus placebo

2. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Description: Summary tables of serious AEs (SAEs) and all other non-serious AEs are located in the Reported Adverse Event Module.
Time Frame: Baseline through end of study (up to 32 months)
Population: The number of participants analyzed was based on the safety population (SP). The SP included participants who received at least 1 dose of enzastaurin or placebo during the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Enzastaurin | Placebo
Number analyzed (Participants) | 24 | 15
Participants
  SAEs | 2 | 0
  Other Non-Serious AEs | 24 | 10

ADVERSE EVENTS:
Arm/Group | Enzastaurin | Placebo
Serious Adverse Events (participants affected / at risk) | 2/24 | 0/15
Other Adverse Events (participants affected / at risk) | 24/24 | 10/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Enzastaurin (N=24) | Placebo (N=15)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Enzastaurin (N=24) | Placebo (N=15)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Conduction disorder (Cardiac disorders) | 0 (0) | 1 (1)
Extrasystoles (Cardiac disorders) | 0 (0) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 2 (2) | 0 (0)
Supraventricular extrasystoles (Cardiac disorders) | 2 (3) | 0 (0)
Hearing impaired (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Eye pain (Eye disorders) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 2 (2) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 4 (4) | 2 (2)
Dry mouth (Gastrointestinal disorders) | 2 (2) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 1 (1)
Fatigue (General disorders) | 1 (1) | 2 (2)
Local swelling (General disorders) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 2 (2) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Viral infection (Infections and infestations) | 0 (0) | 1 (1)
Stress fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 2 (3) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 1 (3)
Blood creatinine increased (Investigations) | 2 (2) | 0 (0)
Electrocardiogram QT prolonged (Investigations) | 3 (5) | 1 (1)
Haemoglobin decreased (Investigations) | 6 (7) | 0 (0)
Haemoglobin increased (Investigations) | 0 (0) | 1 (1)
Urine colour abnormal (Investigations) | 4 (4) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 5 (5) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 8 (13) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 6 (9) | 1 (1)
Dizziness (Nervous system disorders) | 2 (2) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1)
Sleep disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Chromaturia (Renal and urinary disorders) | 2 (2) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 2 (3) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 1 (1)

LIMITATIONS AND CAVEATS:
The planned enrollment for the study was 186 participants, but enrollment was terminated early due to the difficulty of accruing participants once 40 were enrolled into the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days